CLINICAL TRIAL: NCT07076615
Title: The Effect of Dapagliflozin on Patients With Cardiomyopathy
Acronym: Dapagliflozin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: May Mohamed Abdalla (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, May Mohamed Abdalla, Senior teaching assistant, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-73-2024; PO.3.4.1 (Other: Cairo University)
Record Dates: First submitted 2025-04-15; First posted 2025-07-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Decompensated Heart Failure (ADHF)
Keywords: ADHF
MeSH Terms: interventions — dapagliflozin; Diuretics

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups in parallel for the duration of the study.
  Arm A: Receives dapagliflozin (10 mg daily) + standard diuretic therapy
  Arm B: Receives standard diuretic therapy alone
  Each group is treated simultaneously, and outcomes are compared between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind randomized controlled trial. Neither the participants nor the investigators (including care providers and outcome assessors) are aware of the treatment assignments. This masking minimizes bias in treatment administration, patient perception, and outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin + Diuretic (Intervention Group) (Experimental): Participants will receive dapagliflozin 10 mg orally once daily in addition to standard intravenous diuretic therapy.
  Intervention(s):
  Drug: Dapagliflozin (DAPA)
  Dose: 10 mg once daily
  Route: Oral
  Other Name(s): Forxiga
  Drug: Intravenous Diuretic
  Standard care intravenous loop diuretics (e.g., furosemide) according to clinical protocol
  Interventions: Drug: Dapagliflozin (DAPA); Drug: Diuretic
- Active Comparator (Active Comparator): Participants will receive standard intravenous diuretic therapy alone, without dapagliflozin.
  Intervention(s):
  Drug: Intravenous Diuretic
  Standard care intravenous loop diuretics (e.g., furosemide) according to clinical protocol
  Interventions: Drug: Diuretic

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Receives dapagliflozin 10 mg once daily + standard intravenous diuretic therapy
  Arms: Dapagliflozin + Diuretic (Intervention Group)
Drug: Diuretic — Arm B (Control Group): Receives standard intravenous diuretic therapy alone

SUMMARY:
This randomized controlled trial evaluates the efficacy and tolerability of early initiation of dapagliflozin in adult patients hospitalized with acute heart failure (AHF). The study aims to assess the effect of dapagliflozin on pulmonary congestion as measured by lung ultrasound (LUS), length of hospital stay, and cardiac and renal biomarkers. A total of 100 patients will be randomized into two groups: one receiving dapagliflozin plus diuretics and the other receiving diuretics alone. Key outcomes include the reduction of extravascular lung water (assessed by B-lines in LUS), improved diuretic response, changes in NT-proBNP, sST2, CA-125, and NGAL levels, and incidence of acute kidney injury. The study will be conducted at the Cardiology and ICU departments at Kasr Al Ainy Hospital, Cairo University

DETAILED DESCRIPTION:
Acute Heart Failure (AHF) is a life-threatening syndrome and a leading cause of hospitalization worldwide. Effective decongestion during AHF episodes is essential for improving patient outcomes and reducing hospital readmissions. Sodium-glucose co-transporter 2 (SGLT2) inhibitors, particularly dapagliflozin, have shown significant promise in improving cardiovascular outcomes in chronic heart failure; however, their role during acute episodes remains under active investigation.

This prospective, randomized controlled trial aims to assess the efficacy and safety of early dapagliflozin initiation in hospitalized adult patients with AHF, irrespective of diabetes status. A total of 100 patients admitted to the Cardiology and Intensive Care Departments of Kasr Al Ainy Hospital, Cairo University, will be enrolled and randomized (1:1) to either standard diuretic therapy alone or dapagliflozin (10 mg once daily) plus diuretics.

The study's primary endpoint is the degree of pulmonary congestion, evaluated through lung ultrasound (LUS) using an 8-zone scanning protocol and quantification of B-lines. Secondary outcomes include hospital length of stay, diuretic response, changes in cardiac biomarkers (NT-proBNP, sST2, and CA-125), renal biomarker NGAL, and incidence of acute kidney injury.

LUS and echocardiography will be performed by certified intensivists using standardized protocols. Biomarkers will be measured via ELISA kits at three time points: within 24 hours of admission, and at discharge.

The hypothesis is that early use of dapagliflozin in AHF enhances decongestion, improves natriuretic response, and enables earlier hospital discharge without increasing adverse renal or metabolic events.

The results of this study will provide valuable insights into the use of SGLT2 inhibitors during the acute phase of heart failure and may inform future clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Acute heart failure as defined by the 2022 American College of Cardiology/American Heart Association (Heidenreich et al., 2022) or 2021 European Society of Cardiology (McDonagh et al., 2021) guidelines, based on typical symptoms and signs of heart failure requiring hospitalization or emergency department visit
* Elevated natriuretic peptide levels
* Includes heart failure with reduced, mildly reduced, or preserved ejection fraction
* Planned use of intravenous diuretic therapy

Exclusion Criteria:

* Type 1 diabetes mellitus
* Urinary tract or genital infection
* Hypovolemia
* Diabetic ketoacidosis
* Serum glucose < 80 mg/dL at enrollment
* Systolic blood pressure < 90 mmHg at enrollment
* History of hypersensitivity to any SGLT2 inhibitor
* Pregnant or breastfeeding women
* Severe primary valvular lesion requiring intervention
* Severe hepatic impairment (Child-Pugh class C)
* Estimated glomerular filtration rate < 25 mL/min/1.73 m² (by MDRD equation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Effect of Dapagliflozin on Pulmonary Congestion Assessed by Lung Ultrasound (LUS) | Day 1 (Baseline) Day 3 within 24 hours prior to hospital discharge (mean 7 days post-admission)
  To evaluate the effect of dapagliflozin on pulmonary congestion in patients hospitalized with acute heart failure, using lung ultrasound to measure the number of B-lines at defined intervals during hospitalization.

SECONDARY OUTCOMES:
Effect of Dapagliflozin on Hospital Length of Stay | From hospital admission to hospital discharge (an average of 7 days)
  To assess the effect of dapagliflozin on the duration of hospitalization, measured in total days from admission to discharge.
Effect of Dapagliflozin on Renal Biomarker NGAL | Baseline (within 24 hours of admission), and within 24 hours prior to hospital discharge (mean 7 days)
  To assess the effect of dapagliflozin on renal injury using the neutrophil gelatinase-associated lipocalin (NGAL) level in ng/mL as a renal biomarker.
Change in NT-proBNP Levels | Baseline (within 24 hours of admission), and within 24 hours prior to hospital discharge (mean 7 days)
  To assess the change in NT-proBNP levels (pg/mL) in patients receiving dapagliflozin during hospitalization for acute heart failure.
Change in Net Fluid Balance | Day 1, Day 2, and Day 3 of hospitalization
  To determine the net fluid balance (fluid input minus output) (mL per 24 hours) to evaluate diuretic efficiency in patients receiving dapagliflozin.
Incidence of Acute Kidney Injury (AKI) Based on KDIGO Criteria | From admission (Day 1) through hospital discharge (up to 14 days)
  To determine the incidence of acute kidney injury (AKI) according to KDIGO guidelines in patients receiving dapagliflozin during hospitalization.
Change in sST2 Levels | Baseline (within 24 hours of admission), and within 24 hours prior to hospital discharge (mean 7 days)
  To evaluate the effect of dapagliflozin on soluble ST2 (sST2) (ng/mL) concentrations in patients with acute heart failure.
Change in CA-125 Levels | Baseline (within 24 hours of admission), and within 24 hours prior to hospital discharge (mean 7 days)
  To measure the change in CA-125 (Cancer Antigen 125) levels (U/mL) in patients treated with dapagliflozin during hospitalization for acute heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it is undecided whether de-identified individual participant data (IPD), including clinical and laboratory data collected during the study, will be shared with external researchers. A final decision regarding IPD sharing will be made upon study completion, taking into consideration ethical, legal, and regulatory factors.